CLINICAL TRIAL: NCT06886880
Title: Endoscopic Findings in Patients With Upper GIT Bleeding in Assiut University Hospital
Brief Title: Endoscopic Findings in Patients With Upper GIT Bleeding
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ebram Salama Faheim Soliman, Doctor, Assiut University
Other Study IDs: Endoscope in GIT bleeding
Record Dates: First submitted 2025-03-15; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: GIT - Gastrointestinal Tract Hemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Endoscopes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: endoscope — findings in upper GIT Endoscopy

SUMMARY:
This study aims to identify the causes of upper gastrointestinal bleeding through comprehensive evaluation via upper endoscopy in Assiut University Hospital and contribute valuable insights into effective management strategies.

DETAILED DESCRIPTION:
Upper gastrointestinal bleeding (UGIB) is a critical medical situation that arises when there is bleeding proximal to the ligament of Treitz [1]. This condition is a leading cause of morbidity and mortality, with death rates ranging from 5-14% and increasing to over 40% in patients with liver disease[2] Symptoms of UGIB may include anemia, hematemesis, melena, or hematochezia [3].

Neoplasms, arteriovenous malformations, esophageal varices, gastric ulcers, gastric erosions, duodenal ulcers, reflux esophagitis, Mallory-Weiss tears, and fundal varices are causes of UGIB [4].

Current strategies for managing UGIB emphasize early recognition and intervention. Endoscopy is the primary diagnostic and therapeutic modality, allowing for direct visualization of the gastrointestinal tract and enabling interventions such as cauterization, clipping, or band ligation to control bleeding [5]. Recent advancements in endoscopic techniques have improved outcomes by facilitating earlier detection and treatment of UGIB episodes. For instance, the use of hemostatic powders and over-the-scope clips has shown promise in managing refractory cases[6,7].

Endoscopic therapies may have resulted in earlier detection and treatment of UGIB, which could have led to a reduction in the incidence and severity of the condition. Upper GI endoscopy is considered the primary modality for identifying the underlying etiology and administering appropriate therapeutic measures to the patient present with upper GIT bleeding by ligation ,clips, electrocoagulation or by taking biopsies that help in diagnosis. The rationale for this research stems from the need to enhance understanding of UGIB's underlying causes and improve patient outcomes through timely endoscopic intervention. By identifying specific etiologies through upper endoscopy[8,9].

ELIGIBILITY:
Inclusion Criteria:

* Adult patients present with upper GIT bleeding of both gender older than 18 years old

Exclusion Criteria:

* 1- Patients younger than 18 2- Pregnant women 3- patients with end stage disease that not fit for endoscopic intervention

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 2.4.1- Type of the study: Prospective cross-sectional study .
  2.4. 2- Study Setting: Assiut University Hospital , Alraghy Hospital, Endoscopy centre.
  2.4. 3- Study subjects:
  1. Inclusion criteria:
     Adult patients present with upper GIT bleeding of both gender older than 18 years old
  2. Exclusion criteria:
     1. Patients younger than 18
     2. Pregnant women
     3. patients with end stage disease that not fit for endoscopic intervention
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Endoscopic Findings in patients with upper GIT Bleeding | one year
  identify the causes of upper gastrointestinal bleeding through comprehensive evaluation via upper endoscopy in Assuit University Hospital and contribute valuable insights into effective management strategies.

REFERENCES:
- [Background] Elsebaey MA, Elashry H, Elbedewy TA, Elhadidy AA, Esheba NE, Ezat S, Negm MS, Abo-Amer YE, Abgeegy ME, Elsergany HF, Mansour L, Abd-Elsalam S. Predictors of in-hospital mortality in a cohort of elderly Egyptian patients with acute upper gastrointestinal bleeding. Medicine (Baltimore). 2018 Apr;97(16):e0403. doi: 10.1097/MD.0000000000010403. PMID 29668596